CLINICAL TRIAL: NCT02719223
Title: The Effect of On-Line Hemodiafiltration Versus High Flux Hemodialysis on Hemodynamic Parameters in Patients With Intra-Dialytic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0002-16
Record Dates: First submitted 2016-01-30; First posted 2016-03-25 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Intradialytic Hypotension
Keywords: Intradialytic hypotension; hemodynamic parameters; Hemodiafiltration; NICAS device (non-invasive cardiac system)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flux Hemodialysis (Experimental)
  Interventions: Device: NICaS
- OL-HDF (Experimental)
  Interventions: Device: NICaS

INTERVENTIONS:
Device: NICaS — The NICaS is a non invasive device for measuring and calculating of hemodynamic parameters including mean arterial pressure (mm/Hg), cardiac index (l/min/m2) and total peripheral resistance (dynes/sec/cm5).

SUMMARY:
Rationale and objectives

1. Patients on On Line Hemodiafiltration (OL- HDF) are more stable hemodynamically with less Intra Dialytic Hypotension (IDH) episodes compared to conventional hemodialysis (HD). The investigator will follow the hemodynamic parameters during the dialysis sessions (HD and OL-HDF) by using the new non invasive technology, the NICAS device.
2. By switching each patient with IDH from HD to OL- HDF, the investigators will evaluate the hemodynamic parameters and compare the two renal replacement treatment modalities, and prove the superiority of OL-HDF over HD regarding the hemodynamic measures.

DETAILED DESCRIPTION:
Intradialytic hypotension (IDH) or a significant fall in blood pressure (BP) is the most common complication that occurs during hemodialysis (HD) treatment, occurring in up to 20-33% of sessions.

Different mechanisms are involved in the pathogenesis of IDH including acute central hypovolemia, may be precipitated by rapid or excessive ultrafiltration that lead to intravascular volume depletion beyond the level of hemodynamic compensatory response. Other proposed mechanisms of intra vascular depletion are volume shift into the extra-vascular space due to rapid reduction in plasma osmolality, slow and incompatible vascular refilling rate and incorrectly low prescribed dry weight.

Autonomic dysfunction occurs in considerable amount of dialysis patients up to about 50% . This dysfunction reduces the ability to produce an adequate sympathetic response in the setting of acute volume diminution.

Due to the complexity of the dialysis treatment and absence of non- invasive technology, few studies followed the hemodynamic changes which occur during a dialysis session especially during IDH episodes.

OL- HDF is a relatively new method of therapy that allows a larger volume of blood filtration during a single dialysis therapy compared with standard hemodialysis.

Compared to conventional HD treatment, OL-HDF treatment was associated with lower incidence of IDH and better hemodynamic stability.

Bioelectrical impedance analysis is a method for estimating body composition in most of the cases. The Non-Invasive Cardiac System (NICaS) device (non-invasive cardiac system) applies the principle of Whole Body Bio-Impedance and provides continuous data regarding the hemodynamic status (i.e. heart rate, stroke volume, cardiac output, cardiac index, and total peripheral vascular resistance) as well as respiration rate and total body water.

Following the hemodynamic changes, the NICaS device will allow to shed light on the physiological mechanisms underlying the IDH phenomenon and prove the superiority of OL-HDF over regular hemodialysis regarding the hemodynamic measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by IDH during one or more dialytic sessions every week

Exclusion Criteria:

* Patients with recent change in chronic medications, chronic liver disease, recent acute coronary event, cardiac arrhythmias and acute infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The superiority of OL-HDF over regular hemodialysis in decreasing the frequency of intradialytic hypertension episodes. | 5 weeks
Mean arterial pressure (mm/Hg) | 5 weeks
Cardiac index (l/min/m2) | 5 weeks
Total peripheral resistance (dynes/sec/cm5) | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Daugirdas JT. Pathophysiology of dialysis hypotension: an update. Am J Kidney Dis. 2001 Oct;38(4 Suppl 4):S11-7. doi: 10.1053/ajkd.2001.28090. PMID 11602456
- [Result] K/DOQI Workgroup. K/DOQI clinical practice guidelines for cardiovascular disease in dialysis patients. Am J Kidney Dis. 2005 Apr;45(4 Suppl 3):S1-153. No abstract available. PMID 15806502
- [Result] Eknoyan G, Beck GJ, Cheung AK, Daugirdas JT, Greene T, Kusek JW, Allon M, Bailey J, Delmez JA, Depner TA, Dwyer JT, Levey AS, Levin NW, Milford E, Ornt DB, Rocco MV, Schulman G, Schwab SJ, Teehan BP, Toto R; Hemodialysis (HEMO) Study Group. Effect of dialysis dose and membrane flux in maintenance hemodialysis. N Engl J Med. 2002 Dec 19;347(25):2010-9. doi: 10.1056/NEJMoa021583. PMID 12490682
- [Result] Chang TI, Paik J, Greene T, Desai M, Bech F, Cheung AK, Chertow GM. Intradialytic hypotension and vascular access thrombosis. J Am Soc Nephrol. 2011 Aug;22(8):1526-33. doi: 10.1681/ASN.2010101119. PMID 21803971
- [Result] Ronco C, Brendolan A, Milan M, Rodeghiero MP, Zanella M, La Greca G. Impact of biofeedback-induced cardiovascular stability on hemodialysis tolerance and efficiency. Kidney Int. 2000 Aug;58(2):800-8. doi: 10.1046/j.1523-1755.2000.00229.x. PMID 10916105
- [Result] Shoji T, Tsubakihara Y, Fujii M, Imai E. Hemodialysis-associated hypotension as an independent risk factor for two-year mortality in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1212-20. doi: 10.1111/j.1523-1755.2004.00812.x. PMID 15327420
- [Result] Zoccali C, Benedetto FA, Tripepi G, Mallamaci F. Cardiac consequences of hypertension in hemodialysis patients. Semin Dial. 2004 Jul-Aug;17(4):299-303. doi: 10.1111/j.0894-0959.2004.17331.x. PMID 15250922
- [Result] Caplin B, Kumar S, Davenport A. Patients' perspective of haemodialysis-associated symptoms. Nephrol Dial Transplant. 2011 Aug;26(8):2656-63. doi: 10.1093/ndt/gfq763. Epub 2011 Jan 6. PMID 21212166
- [Result] Sands JJ, Usvyat LA, Sullivan T, Segal JH, Zabetakis P, Kotanko P, Maddux FW, Diaz-Buxo JA. Intradialytic hypotension: frequency, sources of variation and correlation with clinical outcome. Hemodial Int. 2014 Apr;18(2):415-22. doi: 10.1111/hdi.12138. Epub 2014 Jan 27. PMID 24467830
- [Result] van der Sande FM, Kooman JP, Leunissen KM. Intradialytic hypotension--new concepts on an old problem. Nephrol Dial Transplant. 2000 Nov;15(11):1746-8. doi: 10.1093/ndt/15.11.1746. No abstract available. PMID 11071958
- [Result] Ewing DJ, Winney R. Autonomic function in patients with chronic renal failure on intermittent haemodialysis. Nephron. 1975;15(6):424-9. doi: 10.1159/000180525. PMID 1196462
- [Result] Lilley JJ, Golden J, Stone RA. Adrenergic regulation of blood pressure in chronic renal failure. J Clin Invest. 1976 May;57(5):1190-200. doi: 10.1172/JCI108387. PMID 1262465
- [Result] Daugirdas JT. Dialysis hypotension: a hemodynamic analysis. Kidney Int. 1991 Feb;39(2):233-46. doi: 10.1038/ki.1991.28. No abstract available. PMID 2002637
- [Result] Santoro A. Cardiovascular dialysis instability and convective therapies. Hemodial Int. 2006 Jan;10 Suppl 1:S51-5. doi: 10.1111/j.1542-4758.2006.01192.x. PMID 16441871